CLINICAL TRIAL: NCT00480480
Title: Long-Term Post- War Adjustment in Bosnian Adolescents, Their Parents and Teachers
Brief Title: Randomized Controlled Trial of the Effectiveness of Group Treatment With War-Exposed Bosnian Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham Young University (Other)
Collaborators: UNICEF (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-261 ASB
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2007-05-31 (Estimated); Status verified 2007-05

CONDITIONS: Posttraumatic Stress Disorder; Depression; Grief (Traumatic Grief and Existential Grief)
Keywords: Trauma; Grief; Depression; Adolescent; War; Group; Therapy; Treatment; Intervention; School; Development
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Prolonged Grief Disorder; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Trauma and Grief Component Therapy for Adolescents (Group Version)

SUMMARY:
Context: This is the first multi-site randomized controlled study of the effectiveness of a group treatment for war-exposed adolescents delivered in-country within a public school system.

Objective: To evaluate the effectiveness of a trauma/grief-focused group treatment program in reducing symptoms of posttraumatic stress disorder (PTSD), depression, and traumatic grief in war-exposed Bosnian youths attending 10 secondary schools located in Central Bosnia.

DETAILED DESCRIPTION:
Design: A randomized controlled trial conducted during the 2000-2001 school year, with 4-month follow-up, compared group treatment to a psychoeducation/skill-based school milieu intervention.

Setting and Participants: Students attending 10 Bosnian secondary schools exposed to severe trauma, traumatic loss, and severe adversity, reporting severe persisting symptoms of PTSD, depression, or traumatic grief, and functional impairment.

Intervention: Students were randomly assigned to either 17-session Trauma and Grief Component Therapy (n=71), or a school milieu intervention (n=73), both conducted by trained school counselors.

ELIGIBILITY:
Inclusion Criteria:

* Significant trauma exposure before, during, or after the war (e.g., serious physical injury, life threat, witnessing death or serious injury, traumatic bereavement);
* Significant current distress, especially severe persisting symptoms of PTSD, depression, or traumatic grief;
* Significant functional impairment in family or peer relationships and school performance

Exclusion Criteria:

* Acute risk status (e.g., suicidal plans and intent)
* Psychosis
* Severe substance abuse (severe enough to interfere with engagement in treatment).

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2000-09; Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
UCLA PTSD Reaction Index | Pre-treatment, post-treatment, and at 4-month follow-up
Depression Self-Rating Scale | Pre-treatment, post-treatment, and 4-month follow-up
UCLA Grief Scale | Pre-treatment, post-treatment

SECONDARY OUTCOMES:
Cognitive Distortions Scale | Pre-treatment and post-treatment
War Exposure Index | Pre-treatment (screening survey)
Post-War Adversities Scale | Pre-treatment (screening survey)
Trauma Reminder Screening Scale | Pre-treatment (screening survey)
Loss Reminder Screening Scale | Pre-treatment (screening survey)
Youth Outcome Questionnaire (Somatic and Interpersonal Problems Subscales) | Pre- and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Layne, Ph.D., Principal Investigator — Brigham Young University, Provo, Utah, USA